CLINICAL TRIAL: NCT05309044
Title: Evaluation of the Efficacy of the Planetary Health Diet Included in an Intensive Lifestyle Change Program on Weight and Body Fat at 4 Months in Mexican Adults With Overweight or Obesity in an Online Modality: Randomized Controlled Trial.
Brief Title: Evaluation of the Planetary Health Diet Included in a Lifestyle Program in Overweight or Obese Mexican Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Doctor, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSP-ONLINE-MX
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Overweight; Obesity
Keywords: Lifestyle intervention; Weight loss; Diet; Planetary health
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Planetary Health Diet Group (Active Comparator): Diet proportional to the EAT-Lancet reference diet, in addition to a behavioral change protocol.
  Interventions: Behavioral: Planetary Health Diet Group
- Low-fat diet group (Active Comparator): Low-fat, low-calorie diet and a behavioral change protocol
  Interventions: Other: Low-fat diet group
- Waiting list group (Placebo Comparator): Waiting list group
  Interventions: Other: Waiting list group

INTERVENTIONS:
Behavioral: Planetary Health Diet Group — This group includes a diet proportional to the EAT-Lancet reference diet (2500 kcal), with a caloric intake of 1200 to 1800 kcal, in addition to a behavioral change protocol during the time of the study (4 months).
  Arms: Planetary Health Diet Group
Other: Low-fat diet group — This group includes a low-fat, low-calorie diet (1200-1800 kcal), in addition to a behavioral change protocol
  Arms: Low-fat diet group
Other: Waiting list group — This group will only receive digital information with recommendations on healthy eating. When the study has finished, this group will receive a behavioral change protocol with a low-fat, low-calorie diet.
  Arms: Waiting list group

SUMMARY:
The EAT-Lancet Commission proposed the planetary health diet as a strategy to achieve health and sustainability goals. Currently, its effect in the treatment of obesity has not been evaluated. The main aim is to evaluate the efficacy of the planetary health diet included in an intensive lifestyle change program compared to a waiting list group, on weight and body fat at 4 months, in Mexican adults with overweight or obesity, in an online modality. This study is a 4-month randomized controlled trial, in an online modality in individuals with overweight or obesity randomly assigned 1:1:1 to one of three groups: 1) planetary health diet, 2) waiting list and 3) low fat-diet. The primary outcome is the difference in change in weight (kg) and body fat (kg) at 4 months between the planetary health diet group and the waiting list group. Comparison with the low-fat diet group will be an exploratory analysis. Secondary variables include changes in waist circumference, BMI, blood pressure, and health-related quality of life. Between group comparisons will be analyzed by intention-to-treat. The protocol was approved by a Research Bioethics Committee.

DETAILED DESCRIPTION:
The present study is a randomized controlled trial of parallel groups and superiority. The sample will consist of 60 participants (20 participants for each arm of the study), calculated from previous studies of our research group. The intervention groups will be 1) planetary health diet, 2) waiting list group, and 3) low-fat diet.

Participants will be measured at the start of the study and at 4 months. The participants of the two diets will follow the Diabetes Prevention Program (DPP) adapted to the Mexican population and its online application. It has also been adapted for the planetary health diet group.

Participants will receive 13 online group educational sessions over 4 months (1 per week) and at least one individual session per week. They will receive a meal plan according to the dietary group to which they belong, with a calorie range from 1200 to 1800 kcal.

Participants in the waiting list group will receive digital information on healthy eating. Upon completion of the study, they will be invited to participate in the "Lifestyle Balance Program" offered at the Nutritional Health Promotion Center, which is an adaptation of the DPP. During the 4 months, there won't be any contact with this group.

The analysis of the primary and secondary outcomes will be carried out in a conservative way by intention to treat and also by completers analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mexican adults (≥18 and ≤60 years).
* Residents of the city of Hermosillo, Sonora.
* BMI ≥ 25 kg/m2 and ≤ 40 kg/m2.
* Availability of time to participate in the study
* Have an electronic device with internet access
* Completion of a dietary record for at least 2 days prior to the intervention.
* Active Facebook account, telephone number, WhatsApp and/or e-mail address
* Basic computer skills

Exclusion Criteria:

* Illiteracy
* Present health conditions due to previous diagnosis with effect on body weight, or that prevent adherence to the intervention (Diabetes, hypertension with values ≥ 150/95 mm Hg, liver failure)
* Pregnancy or lactation.
* History of weight loss in the last 4 months of > 5% of total body weight.
* Being 10% below usual weight.
* Surgeries aimed at weight and/or body fat reduction.
* Use of medications or substances with effect on body weight, e.g. metformin, orlistat, corticosteroids, etc.
* Use of addictive substances
* Plan to change residence during the 4 months of the study.
* Other family member who has agreed to participate in the study.
* History of COVID-19 that required hospitalization or needed for supplemental oxygen or developed sequelae that precludes intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | baseline and 4 months
  To obtain weight (kg), a SECA mBCA model 514 digital scale will be used.
Change in body fat | baseline and 4 months
  Kilograms of total body fat will be obtained by SECA mBCA model 514 digital scale.

SECONDARY OUTCOMES:
Change in waist circumference | baseline and 4 months
  The umbilical scar will be taken as reference and a Lufkin metallic anthropometric tape (Lufkin Executive. Thinline with scale from 0 to 200 cm. Model: W606PMMX) will be used.
Change in the Short Form-36 Health Survey score | baseline and 4 months
  The SF-36 Health Survey evaluates dimensions of health-related quality of life in the adult population (over 16 years of age). It should preferably be self-administered, and it provides eight scales or concepts related to disease and treatment. These scales are: physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health. The SF-36 Health Survey consists of 36 questions (items) that assess both positive and negative health status. The answers to each question are coded and decoded (10 questions), and the result is interpreted on a scale from 0 to 100.
Change in systolic and diastolic blood pressure | baseline and 4 months
  Blood pressure will be measured using an Omron digital blood pressure monitor (model HEM-907XL, Omron Healthcare Co., Ltd, USA). The technique for obtaining blood pressure will be that proposed by the International Society of Hypertension. Three measurements will be taken at 1-minute intervals, and the mean of the last 2 measurements will be used.
Adherence to intervention | up to 16 weeks
  To measure adherence to the interventions, a numerical self-assessment scale from 1 to 5 will be used, where 1 is the lowest score and 5 is the highest, to indicate how adherent they were to the meal plans.
Retention / desertion | 4 months
  The retention percentage will be obtained by dividing the number of people that finished the intervention (i.e. participated in the measurements at 4 months) by the number that started the intervention, multiplied by 100. The dropout percentage will be obtained by the difference in the number of subjects who started and finished the intervention, multiplied by 100.
Change in body mass index | baseline and 4 months
  body mass index is obtained by dividing the weight in kg by the height in meters squared and will be classified in different global BMI cut-off points for adults

CONTACTS AND LOCATIONS:
Overall Officials: Rolando G Diaz Zavala, Ph.D., Principal Investigator — Universidad de Sonora
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The database and results of the study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: Undefined
Access Criteria: Direct communication with the corresponding authors.